CLINICAL TRIAL: NCT02559323
Title: LIVESTRONG Survivorship Care Plan: Continued Data Collection and Follow Up Survey
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 04910
Record Dates: First submitted 2015-08-19; First posted 2015-09-24 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Cancer Patient
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey

SUMMARY:
Cancer survivors face unique health challenges as a result of their cancer diagnosis and treatment. OncoLink created an Internet based program for survivors to learn about their risks. A follow up survey will allow us to continue to develop the program in ways that will benefit users. This survey will need to be conducted via email, which will require the collection of the users email address and a secure method of linking the users care plan questionnaire answers to their survey answers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* 18 years of age and older

Exclusion Criteria:

* Persons who have never had cancer. This program is designed for survivors of adult cancers.
* Survivors of childhood cancers are referred to the Children's Oncology Group Long Term Follow up Guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with cancer diagnosis
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects completing questionnaires | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Metz, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States